CLINICAL TRIAL: NCT05747469
Title: Use of Allograft Adipose Matrix for Small Joint Arthritis of the Hand
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: Musculoskeletal Transplant Foundation (Other)
Responsible Party: Principal Investigator, Meghan McCullough, MD, Principal Investigator, Cedars-Sinai Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00002134
Record Dates: First submitted 2023-02-05; First posted 2023-02-28 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-11

CONDITIONS: Osteoarthritis Hand
MeSH Terms: interventions — Anesthesia, Local; Lidocaine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Adipose Allograft Matrix (AAM) (Other): Using fluoroscopic guidance (X-ray), a needle will be injected into the joint space. 1 cc of Leneva (adipose allograft matrix, MTF Biologics) will be injected into the joint.
  Interventions: Drug: local anaesthetic injection; Procedure: Human Adipose Allograft

INTERVENTIONS:
Drug: local anaesthetic injection — Subcutaneous local anesthesia with 1% lidocaine without epinephrine is administered to the skin overlying the joint.
  Other Names: Lidocaine
Procedure: Human Adipose Allograft — Light axial traction of the digit is used to open the joint space when introducing the 18-gauge needle. Fluoroscopy is used to assist with visualization 1 cc of Leneva is injected into the CMC joint and 0.5 cc in the IP, PIP and DIP joints. The puncture is dressed with a band-aid and coban wrap, which will be worn for 48 hours. Return to work and normal use of the hand is recommended at 48 hours. No narcotics are prescribed.
  Other Names: Leneva

SUMMARY:
The purpose the research is to evaluate the safety and efficacy of injection of adipose allograft matrix (AAM) to the small joints of the hand for treatment of early stage osteoarthritis. The hypothesis is that use of AAM injected directly into the joint will show improvements in pain and disability while providing a safe, off-the-shelf alternative which can obviate the need for, and risks associated with, current treatment options with autologous fat transfer.

As standard of care, routine strength, pain scale scores (VAS) and range of motion will be recorded, a baseline disability survey (DASH score) will also be administered. After these have all been recorded and administered in a separate visit the patient will undergo the lipofilling procedure.

The subject population will include patients over the age of 18 who present with joint pain of the hand with radiographic evidence of osteoarthritis.

DETAILED DESCRIPTION:
The investigators central hypothesis is that use of AAM injected directly into the joint will show improvements in pain and disability while providing a safe, off-the-shelf alternative which can obviate the need for, and risks associated with, current treatment options. The overall aim of the project is to validate the clinical use of AAM for the treatment of early-stage osteoarthritis of the hand in adult patients (>18 years of age). The specific aims for this project are:

1. To determine the safety of use of Leneva as a lipofilling alternative to autologous fat grafting for arthritis of the hand

   a. To determine safety, the investigators will evaluate for any adverse reactions to the injection at each of the follow up time-points
2. To determine the efficacy of the technique as measured by clinical outcomes in terms of pain, disability, range of motion and strength

   a. To determine efficacy, the investigators will measure visual analogue pain scale scores as measures by visual analogue scale, disability scores as measured with DASH scores, and standardized range of motion and strengths scores as measured by the same study administrator at each of the follow up time points
3. To determine patient satisfaction with the procedure a. To determine patient satisfaction, the investigators will administer a survey at each of the follow up time points

ELIGIBILITY:
Inclusion Criteria:

* Patients greater than 18 years, with presentation to the Cedars Sinai hand clinic for joint pain of the hand carpometacarpal, interphalangeal, proximal interphalangeal, and distal interphalangeal joints (CMC, IP, PIP or DIP joints).
* Radiographic evidence of osteoarthritis.

Exclusion Criteria:

* Prior intervention for the presenting joint (either in the form of cortisone or hyaluronic acid injection or surgery).
* Rheumatoid or other inflammatory arthritis condition
* Collagen vascular disease
* Pregnancy or breast-feeding
* Congestive heart failure
* Chronic obstructive pulmonary disease
* Chronic renal failure
* Those who had medication or oral supplements for the previous 4 weeks that could prolong bleeding time (e.g.; Aspirin, Plavix).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2023-08-28 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Range of Motion | Pre-procedure
  Measured with a standardized goniometer
Range of Motion | 6 weeks
  Measured with a standardized goniometer
Range of Motion | 6 month
  Measured with a standardized goniometer
Range of Motion | 12 months
  Measured with a standardized goniometer
Strength Measures | Pre-procedure
  Strength to grip, key pinch and tip pinch, as measured by Jamar dynamometer device)
Strength Measures | 6 weeks
  Strength to grip, key pinch and tip pinch (as measured by Jamar dynamometer device)
Strength Measures | 6 months
  Strength to grip, key pinch and tip pinch (as measured by Jamar dynamometer device)
Strength Measures | 12 months
  Strength to grip, key pinch and tip pinch (as measured by Jamar dynamometer device)
Pain scale scores | Pre-procedure
  Measured using the visual analogue scale (VAS) scored 0 (no pain=better outcome) to 10 (worst pain=worse outcome)
Pain scale scores | 6 weeks
  Measured using the visual analogue scale (VAS) scored 0 (no pain=better outcome) to 10 (worst pain=worse outcome)
Pain scale scores | 6 months
  Measured using the visual analogue scale (VAS) scored 0 (no pain=better outcome) to 10 (worst pain=worse outcome)
Pain scale scores | 12 months
  Measured using the visual analogue scale (VAS) scored 0 (no pain=better outcome) to 10 (worst pain=worse outcome)
Disability Measurement | Pre-procedure
  DASH (Disability of the Arm, Shoulder and Hand) score The DASH is a 30-item self-reported questionnaire in which the response options are presented as 5-point Likert scales. Scores range from 0 (no disability) to 100 (most severe disability). This score was designed be useful in patients with any musculoskeletal disorder of the upper limb.
Disability Measurement | 6 weeks
  DASH (Disability of the Arm, Shoulder and Hand) score The DASH is a 30-item self-reported questionnaire in which the response options are presented as 5-point Likert scales. Scores range from 0 (no disability) to 100 (most severe disability). This score was designed be useful in patients with any musculoskeletal disorder of the upper limb.
Disability Measurement | 6 months
  DASH (Disability of the Arm, Shoulder and Hand) score The DASH is a 30-item self-reported questionnaire in which the response options are presented as 5-point Likert scales. Scores range from 0 (no disability) to 100 (most severe disability). This score was designed be useful in patients with any musculoskeletal disorder of the upper limb.
Disability Measurement | 12 months
  DASH (Disability of the Arm, Shoulder and Hand) score The DASH is a 30-item self-reported questionnaire in which the response options are presented as 5-point Likert scales. Scores range from 0 (no disability) to 100 (most severe disability). This score was designed be useful in patients with any musculoskeletal disorder of the upper limb.
Patient satisfaction | Day of procedure
  Five-point Likert scale (from 1 "strong disagree" to 5 "strongly agree") for the following two survey points: Satisfaction of patient with the procedure and would the patient recommend this procedure to others.
Patient satisfaction | 6 weeks
  Five-point Likert scale (from 1 "strong disagree" to 5 "strongly agree") " for the following two survey points: Satisfaction of patient with the procedure and would the patient recommend this procedure to others.
Patient satisfaction | 6 months
  Five-point Likert scale (from 1 "strong disagree" to 5 "strongly agree") for the following two survey points: Satisfaction of patient with the procedure and would the patient recommend this procedure to others.
Patient satisfaction | 12 months
  Five-point Likert scale (from 1 "strong disagree" to 5 "strongly agree") for the following two survey points: Satisfaction of patient with the procedure and would the patient recommend this procedure to others.

SECONDARY OUTCOMES:
Incidence of Adverse Events | 0-12 months
  Recording of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Meghan McCullough, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

REFERENCES:
- [Background] Heyworth BE, Lee JH, Kim PD, Lipton CB, Strauch RJ, Rosenwasser MP. Hylan versus corticosteroid versus placebo for treatment of basal joint arthritis: a prospective, randomized, double-blinded clinical trial. J Hand Surg Am. 2008 Jan;33(1):40-8. doi: 10.1016/j.jhsa.2007.10.009. PMID 18261664
- [Background] Haas EM, Eisele A, Arnoldi A, Paolini M, Ehrl D, Volkmer E, Giunta RE. One-Year Outcomes of Intraarticular Fat Transplantation for Thumb Carpometacarpal Joint Osteoarthritis: Case Review of 99 Joints. Plast Reconstr Surg. 2020 Jan;145(1):151-159. doi: 10.1097/PRS.0000000000006378. PMID 31592943
- [Background] Holland C, Jaeger L, Smentkowski U, Weber B, Otto C. Septic and aseptic complications of corticosteroid injections: an assessment of 278 cases reviewed by expert commissions and mediation boards from 2005 to 2009. Dtsch Arztebl Int. 2012 Jun;109(24):425-30. doi: 10.3238/arztebl.2012.0425. Epub 2012 Jun 15. PMID 22787504
- [Background] McGarry JG, Daruwalla ZJ. The efficacy, accuracy and complications of corticosteroid injections of the knee joint. Knee Surg Sports Traumatol Arthrosc. 2011 Oct;19(10):1649-54. doi: 10.1007/s00167-010-1380-1. Epub 2011 Jan 11. PMID 21222099
- [Background] Buck-Gramcko D. [Denervation of the wrist joint and interphalageal joints]. Handchirurgie. 1969;1(4):179-81. No abstract available. German. PMID 5409431
- [Background] Lucht U, Vang PS, Munck J. Soft tissue interposition arthroplasty for osteoarthritis of the carpometacarpal joint of the thumb. Acta Orthop Scand. 1980 Oct;51(5):767-71. doi: 10.3109/17453678008990872. PMID 7468170
- [Background] Deb R, Sauerbier M, Rauschmann MA. [History of arthroplasty for finger joints]. Orthopade. 2003 Sep;32(9):770-8. doi: 10.1007/s00132-003-0518-y. German. PMID 14508641
- [Background] Bruser P. [Modified volar plate arthroplasty for posttraumatic and idiopathic osteoarthritis of the metacarpophalangeal and proximal interphalangeal joints]. Orthopade. 2008 Dec;37(12):1180-6. doi: 10.1007/s00132-008-1324-3. German. PMID 18972098
- [Background] Swanson AB. Disabling arthritis at the base of the thumb: treatment by resection of the trapezium and flexible (silicone) implant arthroplasty. J Bone Joint Surg Am. 1972 Apr;54(3):456-71. No abstract available. PMID 5055148
- [Background] Swanson AB. Flexible implant arthroplasty for arthritic finger joints: rationale, technique, and results of treatment. J Bone Joint Surg Am. 1972 Apr;54(3):435-55. No abstract available. PMID 5055146
- [Background] Heers G, Grifka J, Borisch N. [First results after implantation of a pyrocarbon-endoprosthesis in patients with degenerative arthritis]. Z Orthop Ihre Grenzgeb. 2006 Nov-Dec;144(6):609-13. doi: 10.1055/s-2006-955189. German. PMID 17187336
- [Background] IJsselstein CB, van Egmond DB, Hovius SE, van der Meulen JC. Results of small-joint arthrodesis: comparison of Kirschner wire fixation with tension band wire technique. J Hand Surg Am. 1992 Sep;17(5):952-6. doi: 10.1016/0363-5023(92)90476-6. PMID 1401814
- [Background] Herold C, Rennekampff HO, Groddeck R, Allert S. Autologous Fat Transfer for Thumb Carpometacarpal Joint Osteoarthritis: A Prospective Study. Plast Reconstr Surg. 2017 Aug;140(2):327-335. doi: 10.1097/PRS.0000000000003510. PMID 28369017
- [Background] Damia E, Chicharro D, Lopez S, Cuervo B, Rubio M, Sopena JJ, Vilar JM, Carrillo JM. Adipose-Derived Mesenchymal Stem Cells: Are They a Good Therapeutic Strategy for Osteoarthritis? Int J Mol Sci. 2018 Jun 30;19(7):1926. doi: 10.3390/ijms19071926. PMID 29966351
- [Background] Black LL, Gaynor J, Adams C, Dhupa S, Sams AE, Taylor R, Harman S, Gingerich DA, Harman R. Effect of intraarticular injection of autologous adipose-derived mesenchymal stem and regenerative cells on clinical signs of chronic osteoarthritis of the elbow joint in dogs. Vet Ther. 2008 Fall;9(3):192-200. PMID 19003780
- [Background] ter Huurne M, Schelbergen R, Blattes R, Blom A, de Munter W, Grevers LC, Jeanson J, Noel D, Casteilla L, Jorgensen C, van den Berg W, van Lent PL. Antiinflammatory and chondroprotective effects of intraarticular injection of adipose-derived stem cells in experimental osteoarthritis. Arthritis Rheum. 2012 Nov;64(11):3604-13. doi: 10.1002/art.34626. PMID 22961401
- [Background] Zhang L, Wang XY, Zhou PJ, He Z, Yan HZ, Xu DD, Wang Y, Fu WY, Ruan BB, Wang S, Chen HX, Liu QY, Zhang YX, Liu Z, Wang YF. Use of immune modulation by human adipose-derived mesenchymal stem cells to treat experimental arthritis in mice. Am J Transl Res. 2017 May 15;9(5):2595-2607. eCollection 2017. PMID 28560007
- [Background] Wu L, Cai X, Zhang S, Karperien M, Lin Y. Regeneration of articular cartilage by adipose tissue derived mesenchymal stem cells: perspectives from stem cell biology and molecular medicine. J Cell Physiol. 2013 May;228(5):938-44. doi: 10.1002/jcp.24255. PMID 23042088
- [Background] Chiari C, Walzer S, Stelzeneder D, Schreiner M, Windhager R. [Therapeutic utilization of stem cells in orthopedics]. Orthopade. 2017 Dec;46(12):1077-1090. doi: 10.1007/s00132-017-3475-6. German. PMID 28986619
- [Background] Banyard DA, Borad V, Amezcua E, Wirth GA, Evans GR, Widgerow AD. Preparation, Characterization, and Clinical Implications of Human Decellularized Adipose Tissue Extracellular Matrix (hDAM): A Comprehensive Review. Aesthet Surg J. 2016 Mar;36(3):349-57. doi: 10.1093/asj/sjv170. Epub 2015 Sep 1. PMID 26333991
- [Background] Sano H, Orbay H, Terashi H, Hyakusoku H, Ogawa R. Acellular adipose matrix as a natural scaffold for tissue engineering. J Plast Reconstr Aesthet Surg. 2014 Jan;67(1):99-106. doi: 10.1016/j.bjps.2013.08.006. Epub 2013 Sep 12. PMID 24035153
- [Background] Han TT, Toutounji S, Amsden BG, Flynn LE. Adipose-derived stromal cells mediate in vivo adipogenesis, angiogenesis and inflammation in decellularized adipose tissue bioscaffolds. Biomaterials. 2015 Dec;72:125-37. doi: 10.1016/j.biomaterials.2015.08.053. Epub 2015 Aug 31. PMID 26360790
- [Background] Adam Young D, Bajaj V, Christman KL. Award winner for outstanding research in the PhD category, 2014 Society for Biomaterials annual meeting and exposition, Denver, Colorado, April 16-19, 2014: Decellularized adipose matrix hydrogels stimulate in vivo neovascularization and adipose formation. J Biomed Mater Res A. 2014 Jun;102(6):1641-51. doi: 10.1002/jbm.a.35109. Epub 2014 Feb 24. PMID 24510423
- [Background] Kokai LE, Sivak WN, Schilling BK, Karunamurthy A, Egro FM, Schusterman MA, Minteer DM, Simon P, D'Amico RA, Rubin JP. Clinical Evaluation of an Off-the-Shelf Allogeneic Adipose Matrix for Soft Tissue Reconstruction. Plast Reconstr Surg Glob Open. 2020 Jan 27;8(1):e2574. doi: 10.1097/GOX.0000000000002574. eCollection 2020 Jan. PMID 32095393
- [Background] Flynn LE. The use of decellularized adipose tissue to provide an inductive microenvironment for the adipogenic differentiation of human adipose-derived stem cells. Biomaterials. 2010 Jun;31(17):4715-24. doi: 10.1016/j.biomaterials.2010.02.046. Epub 2010 Mar 20. PMID 20304481
- [Background] Choi JS, Kim BS, Kim JY, Kim JD, Choi YC, Yang HJ, Park K, Lee HY, Cho YW. Decellularized extracellular matrix derived from human adipose tissue as a potential scaffold for allograft tissue engineering. J Biomed Mater Res A. 2011 Jun 1;97(3):292-9. doi: 10.1002/jbm.a.33056. Epub 2011 Mar 29. PMID 21448993
- [Background] Brown BN, Freund JM, Han L, Rubin JP, Reing JE, Jeffries EM, Wolf MT, Tottey S, Barnes CA, Ratner BD, Badylak SF. Comparison of three methods for the derivation of a biologic scaffold composed of adipose tissue extracellular matrix. Tissue Eng Part C Methods. 2011 Apr;17(4):411-21. doi: 10.1089/ten.TEC.2010.0342. Epub 2011 Feb 5. PMID 21043998